CLINICAL TRIAL: NCT04808440
Title: Evaluation of Intubation Conditions With the Use of Atracurium After a Fixed Three-minute Delay
Brief Title: Intubation Conditions With Atracurium After Three Minutes
Acronym: CINTROI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201463
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Obesity Female Patients Require General Anaesthesia With Intubation and Atracurium Curarization
Keywords: Tracheal intubation; Atracurium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate intubation conditions with the use of atracurium after a fixed three-minute delay

DETAILED DESCRIPTION:
The recommended dose of a non-depolarizing curare to facilitate tracheal intubation is twice the active dose 95 (the dose that reduces muscle force by 95%). At this dosage, curarization of the laryngeal adductors allowing relaxation and abduction (opening) of the vocal cords is considered certain. With atracurium, the dose for intubation is 0.5 mg.kg-1 and the time to full effect is approximately 3 minutes. With the use of newer hypnotics, there are no data evaluating the conditions for intubation after a fixed time of 3 minutes as with current anesthetic practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult female
* Patient to undergo general anesthesia with intubation for scheduled gynecological surgery
* Patient informed about the study and not opposed to it

Exclusion Criteria:

* Patients with severe and morbid obesity (BMI>35kg/m2)
* Pregnancy
* Patients with difficult intubation
* Allergy to atracurium and to any other drug used.
* Patient under tutorship / curatorship
* Not affiliated with social insurance
* Patient with AME

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, no morbid obesity female patients, without risk factors for difficult tracheal intubation (ref IOT difficile) scheduled for gynaecologic surgery were prospectively included in this observational and monocentric study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Intubation condition | 3 minutes after atracurium injection
  The intubating conditions were evaluated on the basis of the consensus conference on Good Clinical Research Practice in Pharmacodynamic Studies of Neuromuscular Blocking Agents. The score used include the following variables: (1) ease of laryngoscopy, (2) vocal cord position, and (3) reaction to the insertion of the endotracheal tube and the cuff inflation (eg, diaphragmatic movement due to patient cough). Each of these variables was rated as (1) excellent, (2) good, or (3) poor. Intubating conditions were scored as excellent if all variables were excellent; the score was good if at least 1 variable was good and the rest were excellent; the conditions were considered poor if any of the variables was rated poor.
  Evaluation of intubation conditions with the use of atracurium after a fixed three-minute delay

CONTACTS AND LOCATIONS:
Locations (1):
- Service Anesthésie Réanimation Chirurgicale Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debaene B, Beaussier M, Meistelman C, Donati F, Lienhart A. Monitoring the onset of neuromuscular block at the orbicularis oculi can predict good intubating conditions during atracurium-induced neuromuscular block. Anesth Analg. 1995 Feb;80(2):360-3. doi: 10.1097/00000539-199502000-00026. PMID 7818124
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Plaud B, Baillard C, Bourgain JL, Bouroche G, Desplanque L, Devys JM, Fletcher D, Fuchs-Buder T, Lebuffe G, Meistelman C, Motamed C, Raft J, Servin F, Sirieix D, Slim K, Velly L, Verdonk F, Debaene B. Guidelines on muscle relaxants and reversal in anaesthesia. Anaesth Crit Care Pain Med. 2020 Feb;39(1):125-142. doi: 10.1016/j.accpm.2020.01.005. Epub 2020 Jan 8. PMID 31926308
- [Background] Baillard C, Tamrabet C, Ben Abdallah S, Toussaint S, Cheurfa C. Sample size considerations for studies comparing intubating conditions using quantitative monitoring versus a fixed interval during onset of neuromuscular blockade. Anaesth Crit Care Pain Med. 2022 Dec;41(6):101154. doi: 10.1016/j.accpm.2022.101154. Epub 2022 Sep 7. PMID 36087697